CLINICAL TRIAL: NCT01091441
Title: Permanent Observatory of Heart Failure
Acronym: ODIN
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Juilliere, Professor, French Cardiology Society
Other Study IDs: 06302
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Acute Heart Failure
Keywords: therapeutic education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with heart failure: Patients hospitalized for acute heart failure

SUMMARY:
The observatory consists of a row of data collection on a population composed of all patients with heart failure cared for in centers participating in the national education program for patients (named I-CARE) in the form of two groups. Patients who are undergoing a program of therapeutic education track are listed and included in the group of patients educated. Patients who receive no education or only a minimal element for any reason whatsoever are also listed and included in the group of patients who are not educated.

The following of patients will be periodic after their entry in the observatory, up to 2 years of follow up.

DETAILED DESCRIPTION:
The Center for patients with heart failure cared for in a center practicing therapeutic education dedicated to heart failure.

The definition of heart failure selected for inclusion is that recommended by the European Society of Cardiology : presence of at least two signs or symptoms of heart failure (dyspnea, edema of the ankles crackles) at rest or during exercise associated with objective evidence (preferably by echocardiography) of cardiac dysfunction ( systolic and / or diastolic) (resting) and in case of doubt, a response to specific treatment of heart failure.

All patients who are undergoing a program of therapeutic education track are listed and included in the group of patients educated.

All patients who receive no education or only a minimal element for any reason whatsoever are also listed and included in the group of patients who are not educated.

Follow up is done by CRAs at the French Society of Cardiology, by mailing and phone contacts.

ELIGIBILITY:
Inclusion Criteria:

* Patient with heart failure
* Patient supported by a center participating in the I-CARE french program

Exclusion Criteria:

* Refusal by the patient to be listed in an observatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with heart failure in France
  The definition of heart failure selected for inclusion is that recommended by the European Society of Cardiology (The Task Force for the Diagnosis and Treatment of Congestive Heart Failure of the European Society of Cardiology. Eur Heart J 2005; 26: 1115 -- 1140): presence of at least two signs or symptoms of heart failure (dyspnea, edema of the ankles crackles) at rest or during exercise associated with objective evidence (preferably by echocardiography) of cardiac dysfunction ( systolic and / or diastolic) (resting) and in case of doubt, a response to specific treatment of heart failure
Sampling Method: Probability Sample
Enrollment: 3248 (Actual)
Dates: Start 2007-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 2 years
  To analyse survival after 2 years of follow-up (all-causes death)

SECONDARY OUTCOMES:
Recurrence of heart failure | 2 years
  Analyze the data of disease: recurrence of heart failure
Therapeutic | 2 years
  Analyze the data of disease: therapeutic took 2 years of follow-up
Number of participants with adverse events | 2 years
  Analyze the data of disease: cardiovascular events or other non-cardiovascular

CONTACTS AND LOCATIONS:
Locations (1):
- Brabois-Nancy University Hospital, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Result] Schockmel M, Agrinier N, Jourdain P, Alla F, Eicher JC, Coulon P, Druelle J, Mulak G, Danchin N, Thilly N, Juilliere Y; ODIN cohort participants. Socioeconomic factors and mortality in diastolic heart failure. Eur J Clin Invest. 2014 Apr;44(4):372-83. doi: 10.1111/eci.12246. Epub 2014 Feb 19. PMID 24467732
- [Result] Juilliere Y, Suty-Selton C, Riant E, Darracq JP, Dellinger A, Labarre JP, Druelle J, Mulak G, Danchin N, Jourdain P; ODIN cohort participants. Prescription of cardiovascular drugs in the French ODIN cohort of heart failure patients according to age and type of chronic heart failure. Arch Cardiovasc Dis. 2014 Jan;107(1):21-32. doi: 10.1016/j.acvd.2013.11.001. Epub 2013 Dec 30. PMID 24388162
- [Result] Juilliere Y, Jourdain P, Suty-Selton C, Beard T, Berder V, Maitre B, Trochu JN, Drouet E, Pace B, Mulak G, Danchin N; ODIN Cohort Participants. Therapeutic patient education and all-cause mortality in patients with chronic heart failure: a propensity analysis. Int J Cardiol. 2013 Sep 20;168(1):388-95. doi: 10.1016/j.ijcard.2012.09.030. Epub 2012 Oct 6. PMID 23046596
- [Result] Agrinier N, Schockmel M, Thilly N, Laborde-Casterot H, Jourdain P, Alla F, Leclercq C, Dany F, Druelle J, Drouet E, Mulak G, Juilliere Y; ODIN cohort participants. Effectiveness of a patient education programme in heart failure with preserved ejection fraction: Results from the ODIN cohort study using propensity score matching. Arch Cardiovasc Dis. 2018 Jan;111(1):5-16. doi: 10.1016/j.acvd.2017.03.010. Epub 2017 Sep 22. PMID 28943262
- [Result] Garbacz L, Juilliere Y, Alla F, Jourdain P, Guyon G, Coudane H, Herve C, Claudot F. Perception of therapeutic patient education in heart failure by healthcare providers. Arch Cardiovasc Dis. 2015 Aug-Sep;108(8-9):446-52. doi: 10.1016/j.acvd.2015.03.008. Epub 2015 Jun 10. PMID 26071349